CLINICAL TRIAL: NCT06925763
Title: Unlocking the Regenerative Potential: The Effect of Nitroglycerin Hydrogel on Repairing Critical Bone Defects (Experimental Study)
Brief Title: Effect of Nitroglycerin Hydrogel on Repairing Critical Bone Defects
Acronym: Nitro- Bone
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Minia University (Other)
Responsible Party: Principal Investigator, shaimaa hamdy, Dr Shaimaa Hamdy principal investigator, Minia University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Nitroglycerin bone healing; ethical committee no. 108 (Other: ethical committee no. 108)
Record Dates: First submitted 2025-04-07; First posted 2025-04-13 (Actual); Last update posted 2025-04-13 (Actual); Status verified 2025-01

CONDITIONS: Bone Regeneration; Periodontal Bone Loss; Healing Fracture of Bone
Keywords: nitroglycerin,; bone regeneration; critical size defect
MeSH Terms: conditions — Alveolar Bone Loss | interventions — Nitroglycerin

STUDY DESIGN:
Intervention Model Description: All the animals were adult, ranging in age from 3 to 7 months and in weight between 250 and 350 g.
  The control group: was filled with a placebo hydrogel negative control. while the study group 1: was filled with 30 μM Nitroglycerin-loaded hydrogel positive control.
  Study group 2: was filled with 50 μM Nitroglycerin-loaded hydrogel positive control.
  thirty-three rats will be sacrificed after two weeks, and the others will be saved.
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- control group (Placebo Comparator)
  Interventions: Drug: Nitroglycerin
- the study group 1 (Experimental): was filled with 30 μM Nitroglycerin-loaded hydrogel (positive control)
  Interventions: Drug: Nitroglycerin
- Study group 2 (Experimental): was filled with 50 μM Nitroglycerin-loaded hydrogel (positive control).
  Interventions: Drug: Nitroglycerin

INTERVENTIONS:
Drug: Nitroglycerin — cardiac disease treatment drug

SUMMARY:
Due to their osteoconductive, osteoinductive, and osteogenic qualities, autologous bone grafts are the gold standard for augmenting bone, (1). However, problems, insufficient bone quantity, and/ or quality at the donor location could prevent it from being used. Consequently, a variety of bone graft materials, such as allografts and/or xenografts, were developed to improve bone development and provide an osteoconductive matrix in the so-called hard tissue critical-size defect (CSD) (2).

"critically-sized" defect is regarded as one that would not heal spontaneously despite surgical stabilization and requires further surgical intervention (3). The management of critical-sized bone defects remains a major clinical orthopedic challenge. Critical-sized bone defects are technically defined as those that will not heal spontaneously during the patient's lifetime. Bone loss greater than 2 times the diameter of the long bone diaphysis is unlikely to result in union despite appropriate stabilization methods (4).

Nitroglycerin, also known as glyceryl trinitrate (GTN), is a medication commonly used to treat heart conditions like angina pectoris and chronic heart failure. It acts as a potent vasodilator, dilating the vascular system to improve blood flow. Nitroglycerin has been found to have a positive effect on bone formation. Studies indicate that Nitroglycerin when applied topically, can increase bone formation and reduce bone resorption. This effect is achieved through the stimulation of osteoblastic differentiation and proliferation (5).

The mechanism of action of Nitroglycerin in bone formation involves its conversion into nitric oxide (NO), which plays a crucial role in stimulating bone formation. Nitric oxide released from nitroglycerin acts as a signaling molecule that enhances osteoblastic differentiation and proliferation of bone marrow-derived mesenchymal stem cells. This process leads to increased bone mineral density, improved bone geometry, and enhanced bone strength (5).

Hydrogels are natural or synthetic biocompatible polymers that are widely used in periodontal tissue engineering as a delivery material for different biologics (6). Synthetic hydrogels have superiority in chemical and mechanical properties over natural hydrogels (7). Carbopol or polyacrylic acid (PAA) is one of the most widely used polymers as a hydrogel. It is an anionic polyelectrolyte that can be readily polymerized and crosslinked to form hydrogels with a swelling capacity greater than their dry weight (8).

DETAILED DESCRIPTION:
Aim of the study Histomorphometric analysis of Regenerative Capacity of Nitroglycerin-loaded hydrogel in management of critical size bone defect in Experimental study.

Materials and Methods

ELIGIBILITY:
Inclusion Criteria:

* All animals were adult with an age ranging between 3 to 7 months and a weight ranging between 250 and 350 g

Exclusion Criteria:

* other than inclusion

Max Age: 7 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Gender Based: Yes
Enrollment: 33 (Estimated)
Dates: Start 2025-04-01 (Estimated); Primary Completion 2025-04-03 (Estimated); Study Completion 2025-08-01 (Estimated)

PRIMARY OUTCOMES:
radiographic analysis | baseline, 2months
  bone formation in the critical size was evaluated by radiographic measurements

CONTACTS AND LOCATIONS:
Locations (1):
- Shaimaa Hamdy, Cairo, Cairo- Egypt, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rodriguez-Eguren A, Bueno-Fernandez C, Gomez-Alvarez M, Frances-Herrero E, Pellicer A, Bellver J, Seli E, Cervello I. Evolution of biotechnological advances and regenerative therapies for endometrial disorders: a systematic review. Hum Reprod Update. 2024 Oct 1;30(5):584-613. doi: 10.1093/humupd/dmae013. PMID 38796750
- See also: Nitroglycerin in bone regeneration — https://pubmed.ncbi.nlm.nih.gov/?term=nitroglycerin+in+bone+regeneration
- Available data/document: Individual Participant Data Set — https://pubmed.ncbi.nlm.nih.gov/?term=nitroglycerin+in+bone+regeneration